CLINICAL TRIAL: NCT06971094
Title: A Multicenter, Randomized, Open-Label, Standard-of-Care-Controlled, Phase III Clinical Trial to Evaluate the Safety and Efficacy of Intrathecal (IT) Injection of GC101 Adeno-Associated Virus Injection in the Treatment of Patients With Type 2 Spinal Muscular Atrophy (SMA)
Brief Title: Safety and Efficacy Evaluation of GC101 Gene Therapy Via Intrathecal (IT) Injectionin the Treatment of Patients With Type 2 Spinal Muscular Atrophy (SMA) - Phase III
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC101-SMA-011
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: SMA - Spinal Muscular Atrophy
Keywords: SMA, type II, AAV gene therapy; Genecradle
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: This trial employs a multicenter, randomized, open-label, standard-of-care-controlled design and plans to enroll 50 patients with Type 2 SMA aged 2 to 12 years who have previously received treatment. The trial consists of two groups: one group will receive a single intrathecal injection of GC101 at a dose of 1.2E+14 vg per person and discontinue their previous standard-of-care treatment with nusinersen; the other group will continue their previous standard-of-care treatment with nusinersen. Participants will be randomly assigned to the trial group or the control group in a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC101 (Experimental): single dose of GC101 at dosage of 1.2E+14 vg per person via intrathecal injection
  Interventions: Genetic: GC101 adeno-associated virus injection
- Control (No Intervention): Participants will continue to receive treatment according to their previous standard-of-care regimen with nusinersen.

INTERVENTIONS:
Genetic: GC101 adeno-associated virus injection — Self-complementary recombinant adeno-associated viral vector (scAAV) containing a single-stranded transgene encoding a codon-optimized human SMN1 gene
  Arms: GC101

SUMMARY:
This trial employs a multicenter, randomized, open-label, standard-of-care-controlled design and plans to enroll 50 patients with Type 2 SMA aged 2 to 12 years who have previously received nusinersen. The primary objective of the trial is to evaluate the efficacy of GC101 in treating Type 2 SMA. The secondary objectives are to assess the efficacy, safety, and pharmacokinetic (PK) profile of GC101 in treating Type 2 SMA.

DETAILED DESCRIPTION:
The trial is divided into two groups: one group will receive a single intrathecal injection of GC101 at a dose of 1.2E+14 vg per person and discontinue their previous standard-of-care treatment with nusinersen; the other group will continue their previous standard-of-care treatment with nusinersen. Participants will be randomly assigned to the trial group or the control group in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Type 2 5q-SMA through clinical phenotype and genetic testing.
* Patients who have been receiving regular treatment with nusinersen for more than one year prior to screening.
* Patients who have not received treatment with risdiplam within 2 months prior to screening and have no plans to receive risdiplam treatment within 12 months after enrollment.
* Patients who can sit independently but cannot walk independently at the time of screening (according to the definitions of independent sitting and walking in the WHO-MGRS motor milestones scale), and have an HFMSE score of ≥10 points.
* Patients and/or their legal guardians are able to understand and are willing to comply with the requirements and procedures of the trial protocol, and voluntarily participate and sign the informed consent form

Exclusion Criteria:

* Patients with serum anti-AAV9 neutralizing antibody titers > 1:50 at the time of screening.
* Patients who have received nusinersen treatment within 2 months prior to enrollment.
* Patients with any medical conditions that may affect the interpretation of study results or pose a risk to the safety of the participants, including but not limited to organ dysfunction of any cause, acute infectious diseases, primary/acquired immunodeficiency diseases, severe cardiovascular/cerebrovascular diseases, gastrointestinal diseases, diabetes, known epilepsy, meningitis, seizure or convulsion history, or a family history of psychiatric disorders; and those with cerebrospinal fluid circulation disorders.
* Patients with severe liver injury/hepatic insufficiency of any cause, including but not limited to alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≥3 times the upper limit of normal (ULN); total bilirubin (TBil) ≥1.5 times the ULN.
* Patients deemed by the investigator to have contraindications to glucocorticoid use, such as severe hypertension, diabetes, systemic infectious diseases, fungal infections, glaucoma, osteoporosis, peptic ulcer disease, tuberculosis, etc.
* Patients with contraindications to lumbar puncture or intrathecal injection therapy.
* Patients with any medical conditions that may affect the assessment of motor function, such as severe scoliosis, severe joint contracture deformities, planned spinal correction surgery during the trial period, severe osteoporosis, or a history of fractures.
* Patients positive for hepatitis B surface antigen (HBsAg), human immunodeficiency virus (HIV) antibodies, hepatitis C virus (HCV) antibodies, or syphilis antibodies.
* Patients who have received vaccinations within 2 weeks prior to dosing.
* Patients who have previously received gene therapy or participated in any clinical trial within 3 months prior to screening.
* Patients deemed by the investigator to be unsuitable for participation in this study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HFMSE score change from baseline | 52 weeks
  HFMSE Motor Function Assessment (Hammersmith Functional Motor Scale Expanded) is a standardized tool specifically designed to evaluate motor function in patients with spinal muscular atrophy (SMA). It includes 33 test items covering actions such as head control, sitting, standing, walking, stair climbing, jumping, as well as balance and coordination, providing a comprehensive assessment of motor function in the trunk and limbs. The maximum total score is 66 points, with higher scores indicating better motor capabilities.

SECONDARY OUTCOMES:
HFMSE score change from baseline | 26 weeks
The proportion of participants with an increase in HFMSE score of ≥3 points from baseline. | 26 and 52 weeks
  Minimal clinically important differences (MCID) were defined as an HFMSE score improvement of ≥3 points.
Changes in WHO-MGRS motor milestones from baseline. | 26 and 52 weeks
  WHO-MGRS (World Health Organization Multicenter Growth Reference Study) motor development milestones include:
  Sitting without support Standing with support Crawling on hands and knees Walking with support Standing alone Walking alone
RULM score change from baseline. | 26 and 52 weeks
  RULM Motor Function Assessment (Revised Upper Limb Module) is a standardized tool designed to evaluate upper limb function in patients with spinal muscular atrophy (SMA). A maximum total score is 37 points. Higher scores indicate better upper limb performance.
SMAIS score change from baseline. | 26 and 52 weeks
  Spinal Muscular Atrophy Independence Scale （SMAIS）is a patient- and caregiver-reported outcome measure designed to assess the level of assistance required by individuals with Type 2 and non-ambulant Type 3 spinal muscular atrophy (SMA) to perform activities of daily living. Higher scores indicate greater independence, with a range from 0 to 44
The incidence of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs). | 52 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The Seventh Medical Center of Chinese PLA General Hospital, Beijing
  - Children's Medical Center of Peking University First Hospital, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - National Children's Medical Center，Shanghai Jiaotong University, Shanghai
  - Shenzhen Children's Hospital, Shenzhen
  - Children's Hospital of Soochow University, Suzhou
  - Wuhan Children's Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided